CLINICAL TRIAL: NCT06953999
Title: A Randomized, Controlled, Multi-center Phase III Clinical Study of Ivonescimab Plus Chemotherapy With or Without AK117 Versus Placebo Combined With Chemotherapy as First-line Treatment for Metastatic Pancreatic Cancer
Brief Title: A Phase III Study of Ivonescimab + Chemo With/Without AK117 vs Chemo in Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-310
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ivonescimab + AK117 + Albumin-bound Paclitaxel + Gemcitabine (Experimental)
  Interventions: Drug: Ivonescimab, AK117, Albumin-bound Paclitaxel, Gemcitabine
- Ivonescimab + AK117 Placebo + Albumin-bound Paclitaxel + Gemcitabine (Experimental)
  Interventions: Drug: Ivonescimab, AK117 Placebo, Albumin-bound Paclitaxel, Gemcitabine
- Ivonescimab Placebo + AK117 Placebo + Albumin-bound Paclitaxel + Gemcitabine (Active Comparator)
  Interventions: Drug: Ivonescimab Placebo, AK117 Placebo, Albumin-bound Paclitaxel, Gemcitabine

INTERVENTIONS:
Drug: Ivonescimab, AK117, Albumin-bound Paclitaxel, Gemcitabine — Ivonescimab: a specified dose and frequency administrated by intravenous infusion (IV).
  AK117: a specified dose and frequency administrated by intravenous infusion (IV).
  Albumin-bound Paclitaxel: 125 mg/m2 weekly for 3 weeks followed by 1 week of rest.
  Gemcitabine: 1000 mg/m2 weekly for 3 weeks followed by 1 week of rest.
  Arms: Ivonescimab + AK117 + Albumin-bound Paclitaxel + Gemcitabine
Drug: Ivonescimab, AK117 Placebo, Albumin-bound Paclitaxel, Gemcitabine — Ivonescimab: a specified dose and frequency administrated by intravenous infusion (IV).
  AK117 Placebo: a specified dose and frequency administrated by intravenous infusion (IV).
  Albumin-bound Paclitaxel: 125 mg/m2 weekly for 3 weeks followed by 1 week of rest.
  Gemcitabine: 1000 mg/m2 weekly for 3 weeks followed by 1 week of rest.
  Arms: Ivonescimab + AK117 Placebo + Albumin-bound Paclitaxel + Gemcitabine
Drug: Ivonescimab Placebo, AK117 Placebo, Albumin-bound Paclitaxel, Gemcitabine — Ivonescimab Placebo : a specified dose and frequency administrated by intravenous infusion (IV).
  AK117 Placebo : a specified dose and frequency administrated by intravenous infusion (IV).
  Albumin-bound Paclitaxel: 125 mg/m2 weekly for 3 weeks followed by 1 week of rest.
  Gemcitabine: 1000 mg/m2 weekly for 3 weeks followed by 1 week of rest.
  Arms: Ivonescimab Placebo + AK117 Placebo + Albumin-bound Paclitaxel + Gemcitabine

SUMMARY:
This is a Phase 3, randomized, double-blind clinical trial aimed at evaluating the efficacy and safety of Ivonescimab plus chemotherapy with or without AK117 versus placebo plus chemotherapy in patients with metastatic pancreatic cancer. The study seeks to determine whether the addition of Ivonescimab and/or AK117 improves clinical outcomes compared to standard chemotherapy alone. Participants will be randomly assigned to receive either Ivonescimab with/without AK117 or placebo, both in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form.
2. Age at enrollment is ≥ 18 and ≤ 75 years, both males and females are eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 3 months.
5. Histologically or cytologically confirmed, unresectable metastatic pancreatic ductal adenocarcinoma (PDAC).
6. No prior systemic anti-cancer treatment for metastatic PDAC.
7. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
8. Adequate organ function.

Exclusion Criteria:

1. Histologically or cytologically confirmed other types of pancreatic malignancies or mixed histology types.
2. Presence of active central nerve system (CNS) metastases.
3. Known germline BRCA1/2 or PALB2 mutations.
4. Clinically significant or recurrent pleural effusion, pericardial effusion, or ascites requiring drainage.
5. History of other malignancies within the past 5 years.
6. History of significant bleeding tendencies or coagulopathy; clinically significant bleeding events within 1 month before the first dose.
7. Previous anti-angiogenic therapy and immunotherapy.
8. Active autoimmune disease requiring systemic treatment within the past 2 years.
9. Pregnant or breastfeeding women.
10. Concurrent participation in another clinical trial, unless it is an observational or non-interventional study or in the follow-up phase of an interventional study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 999 (Estimated)
Dates: Start 2025-05-14 (Estimated); Primary Completion 2027-05-14 (Estimated); Study Completion 2028-05-14 (Estimated)

PRIMARY OUTCOMES:
Overall response (OS) | Up to approximately 2 years
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented disease progression (per RECIST v1.1 criteria) assessed by investigators or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , assessed by investigators based on RECIST v1.1.
Disease Control Rate (DCR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1.
Duration of response (DoR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Duration of response (DoR) assessed according to RECIST v1.1.
Time to response (TTR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Time to response (TTR) is defined as the time to response based on RECIST v1.1.
Adverse Events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporarily associated with the use of study treatment, whether or not considered related to the study treatment.
Cmax and Cmin | Up to approximately 2 years
  AK112 serum drug concentrations in subjects at different time points after AK112 administration.
Anti-drug antibodies (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No